CLINICAL TRIAL: NCT03987581
Title: Cost Effectiveness of Combined Contingency Management and Cognitive Behavioral Therapy for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PRO00101744
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Drinking; Veterans
MeSH Terms: conditions — Alcohol Drinking | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBT + mCM + incentive (Experimental): Participants in this arm will receive 12 sessions of cognitive behavioral treatment, mobile contingency management for alcohol abstinence, and a monetary incentive for 30-day abstinence at the 6-month follow-up.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Mobile Contingency Management (mCM); Behavioral: Long-term incentive
- CBT + mCM + no incentive (Experimental): Participants in this arm will receive 12 sessions of cognitive behavioral treatment and mobile contingency management for alcohol abstinence. They will not receive monetary incentive for 30-day abstinence at the 6-month follow-up.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Mobile Contingency Management (mCM)
- CBT alone + incentive (Experimental): Participants in this arm will receive 12 sessions of cognitive behavioral treatment and a monetary incentive for 30-day abstinence at the 6-month follow-up. They will not receive contingency management for alcohol abstinence during the treatment period.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Long-term incentive
- CBT alone + no incentive (Active Comparator): Participants in this arm will receive 12 sessions of cognitive behavioral treatment. They will not receive monetary incentive for 30-day abstinence at the 6-month follow-up. They will not receive contingency management for alcohol abstinence during the treatment period.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Twelve in-person counseling sessions designed to assist participants with becoming abstinent from alcohol use (or reduce use).
  Other Names: CBT
Behavioral: Mobile Contingency Management (mCM) — Abstinence (measured by breath alcohol) will be intermittently reinforced. For each breath alcohol concentration reading that tests negative, a participant will earn a virtual scratch-off lottery ticket that contains 100 different values.
  Other Names: mCM; CM
  Arms: CBT + mCM + incentive; CBT + mCM + no incentive
Behavioral: Long-term incentive — This incentive is $300 for self-reported and bioverified 30-day abstinence from heavy drinking at the follow-up scheduled for 6-months after the initial quit date
  Other Names: Incentive
  Arms: CBT + mCM + incentive; CBT alone + incentive

SUMMARY:
Alcohol contributes to 88,000 deaths and costs an estimated $223 billion annually in the United States. Alcohol use disorder (AUD) is highly prevalent in veterans. The positive public health impact of reducing heavy drinking among veterans with AUD would prevent significant medical morbidity and mortality. Contingency management (CM) is an intensive behavioral therapy that provides incentives to individuals for reducing substance use. Monitoring alcohol abstinence usually requires daily monitoring. Because of this difficulty, CM approaches for treatment of AUD are not currently available to people with AUD. Our group has developed a mobile smart-phone application that allows patients to video themselves using an alcohol breath monitor and transmit the encrypted data to a secure server. This innovation has made the use of CM for outpatient AUD treatment feasible. The aim of the current study is to evaluate the effectiveness and cost effectiveness of CM as an add-on to cognitive behavioral therapy for AUD. The trial will also explore the potential usefulness of a long-term abstinence incentive ontreatment utilization and alcohol outcomes. Proposed is a trial in which 140 veterans with AUD will be randomized to receive either CM as an add-on to evidence-based CBT or CBT alone. Veterans will also be randomized to one of two long-term incentive conditions (i.e., receipt of a monetary incentive for abstinence/low-risk drinking at 6- months vs. no incentive). This project aims to advance AUD treatment by 1) testing the effectiveness of a mobile health approach that makes CM for AUD feasible, and 2) providing highly needed cost-effectiveness data on the use of behavioral incentives as an adjunct to CBT for the treatment of AUD. These aims are designed to address two significant barriers to the implementation of CM for AUD.

ELIGIBILITY:
Inclusion Criteria:

* are an enrolled veteran at the DVAHCS for primary care,
* have current AUD (meeting past month DSM-5 criteria), and
* are willing to make a quit attempt and/or reduce alcohol use to low risk levels.

Exclusion Criteria:

* have fewer than 3 days of abstinence,
* have a history of clinically significant alcohol withdrawal, as indicated by a score of 10 or more on the Clinical Institute Withdrawal Assessment of Alcohol (CIWA), or
* are currently receiving professional behavioral treatment for AUD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven participants were deemed eligible to participate in the study but were not randomized. Seven voluntarily withdrew, and four were lost to contact.
Period: Overall Study
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Started | 35 | 35 | 35 | 35
Completed | 35 | 35 | 35 | 35
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive | Total
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 49 (14) | 50 (15) | 50 (12) | 49 (13)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 29 | 27 | 28 | 28 | 112
  Sex: Female | 6 | 7 | 7 | 7 | 27
  Sex: Unknown, not reported | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 2 | 8
  Not Hispanic or Latino | 32 | 35 | 32 | 33 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 12 | 21 | 15 | 65
  White | 18 | 22 | 12 | 17 | 69
  More than one race | 0 | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 35 | 35 | 140

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Heavy Drinking Days
Description: At the 6-month follow-up visit, participants will self-report the number of heavy drinking (> 5 drinks in day for men, > 4 drinks in a day for women) days they have had in the past thirty days.
Time Frame: 6-month post quit visit
Population: Sixteen participants were excluded from analyses because they were withdrawn or lost to contact prior to the 6-month follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 34 | 30 | 32 | 27
days | 15.1 (12.2) | 15.9 (10) | 13.2 (11.2) | 11.3 (11.2)

2. Secondary Outcome: Average Number of Heavy Drinking Days
Description: At the 12-month follow-up visit, participants will self-report the number of heavy drinking (> 5 drinks in day for men, > 4 drinks in a day for women) days in the past thirty days.
Time Frame: 12-month post quit visit
Population: Thirty-two participants were excluded from analyses because they were withdrawn or lost to contact prior to the 12-month follow-up visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 30 | 26 | 29 | 23
days | 2.8 (7) | 1.2 (3.1) | 2.4 (6.5) | 4.5 (10.4)

3. Secondary Outcome: Average Number of Binge Drinking Days
Description: Participants will self-report the number of binge drinking (heavy drinking within a 2-hour period) days in the past thirty days.
Time Frame: 6-month post quit visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 34 | 30 | 32 | 27
days | 0.9 (4.8) | 3.4 (7.6) | 1.8 (6.5) | 2.2 (6.7)

4. Secondary Outcome: Average Number of Binge Drinking Days
Description: as for outcome 3
Time Frame: 12-month post quit visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 30 | 26 | 29 | 23
days | 0.5 (1.5) | 0.7 (2.8) | 0.8 (3.4) | 4.0 (10.5)

5. Secondary Outcome: Average Number of Drinking Days
Description: Participants will self-report the number of drinking days in the past thirty days.
Time Frame: 6-month post quit visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 34 | 30 | 32 | 27
days | 11.0 (10.2) | 12.2 (11.6) | 7.9 (9.3) | 9.6 (10.7)

6. Secondary Outcome: Average Number of Drinking Days
Description: Participants will self-report the number of drinking days in the past thirty days.
Time Frame: 12-month post quit visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 30 | 26 | 29 | 23
days | 10.5 (10.4) | 8.0 (9.8) | 8.1 (9.9) | 12.3 (11.0)

7. Secondary Outcome: Average Number of Drinks Per Drinking Day
Description: Participants will self-report the number of drinks on drinking days in the past 30 days.
Time Frame: 6-month post quit visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 34 | 30 | 32 | 27
drinks | 3.4 (3.8) | 3.2 (3.3) | 2.5 (2.0) | 2.0 (2.1)

8. Secondary Outcome: Average Number of Drinks Per Drinking Day
Description: Participants will self-report the number of drinks on drinking days in the past 30 days.
Time Frame: 12-month post quit visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 30 | 26 | 29 | 23
drinks | 3.5 (3.7) | 2.3 (2.5) | 3.2 (2.8) | 2.8 (2.0)

9. Secondary Outcome: Number of Participants With Self-reported Abstinence
Description: Participants will self-report whether or not consumed any alcohol in the past 30 days.
Time Frame: 6-month post quit visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 34 | 30 | 32 | 27
Participants | 5 | 6 | 10 | 5

10. Secondary Outcome: Number of Participants With Self-reported Abstinence
Description: Participants will self-report whether or not consumed any alcohol in the past 30 days.
Time Frame: 12-month post quit visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 30 | 26 | 29 | 23
Participants | 5 | 8 | 5 | 3

11. Secondary Outcome: Number of Participants With Bioverification of Low-risk Drinking
Description: Participants will provide a fingerstick blood sample. Phosphatidylethanol (PEth) testing will provide any evidence of excessive alcohol use in previous 4 weeks.
Time Frame: 6-month post quit visit
Population: Sixteen participants were excluded from analyses because they were withdrawn or lost to contact prior to the 6-month follow-up visit. Additionally, 7 participants failed to send in their PEth test kits for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 31 | 30 | 28 | 28
Participants | 13 | 7 | 13 | 9

12. Secondary Outcome: Number of Participants With Bioverification of Low-risk Drinking
Description: as for outcome 11
Time Frame: 12-month post quit visit
Population: Thirty-two participants were excluded from analyses because they were withdrawn or lost to contact prior to the 12-month follow-up visit. Additionally, 4 participants failed to send in their PEth test kits for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 25 | 26 | 29 | 24
Participants | 4 | 13 | 9 | 6

13. Secondary Outcome: Treatment Utilization as Measured by Number of Treatment Visits
Description: Participants will provide self-report on use of adjunct treatments (e.g., Alcoholics Anonymous, group counseling) for alcohol use during the period between post-treatment and follow-ups. Where available, Department of Veterans Affairs administrative data will be used to determine enrollment or involvement in aftercare treatment.
Time Frame: 6-month post quit visit
Population: 29 participants were withdrawn from analyses due to missing data.
Measure: Mean (Standard Deviation); unit: treatment visits
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 29 | 27 | 29 | 26
treatment visits | 0.03 (0.2) | 1.5 (4.5) | 2.1 (5.2) | 0.2 (0.7)

14. Secondary Outcome: Treatment Utilization as Measured by Number of Treatment Visits
Description: as for outcome 13
Time Frame: 12-month post quit visit
Population: 31 participants were withdrawn from analyses due to missing data.
Measure: Mean (Standard Deviation); unit: treatment visits
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 28 | 25 | 31 | 25
treatment visits | 0.6 (1.6) | 8.2 (29.5) | 2.9 (8.9) | 0.3 (1.0)

15. Secondary Outcome: Health Care Related Quality of Life
Description: Health care related quality of life will be measured by the EuroQol.
Time Frame: 12-month post quit visit
Reporting Status: Not Posted

16. Secondary Outcome: CBT Treatment Engagement as Measured by the Number of Cognitive Behavioral Therapy Treatment Sessions Completed
Description: The number of cognitive behavioral therapy treatment sessions completed by each participant will be measured to determine treatment engagement
Time Frame: Post-treatment, approximately 14 weeks
Population: Two participants were withdrawn from analyses due to missing data.
Measure: Mean (Standard Deviation); unit: CBT sessions
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
Number analyzed (Participants) | 35 | 35 | 35 | 33
CBT sessions | 10.4 (2.9) | 9.6 (3.3) | 9.1 (3.8) | 9.3 (3.9)

17. Secondary Outcome: Incremental Cost-Effectiveness Ratio
Description: Measure of cost-effectiveness; costs as the numerator and effectiveness as measured by quality-adjusted life years (QALY) as the denominator
Time Frame: 12-month post quit visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to one-year follow-up (about one year)
Arm/Group | CBT + mCM + Incentive | CBT + mCM + no Incentive | CBT Alone + Incentive | CBT Alone + no Incentive
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 4/35 | 3/35 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT + mCM + Incentive (N=35) | CBT + mCM + no Incentive (N=35) | CBT Alone + Incentive (N=35) | CBT Alone + no Incentive (N=35)
increase in psychological distress (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2) — Increase in psychiatric distress due to participating in interviews and completing questionnaires related to symptoms.
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — headache due to alcohol withdrawal
frustration (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — frustration with technology used in study
irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — irritability due to alcohol withdrawal
nightmares (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — nightmares about alcohol use after a period of abstinence
abnormal skin sensations (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — abnormal skin sensations due to alcohol withdrawal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03987581/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03987581/ICF_001.pdf